CLINICAL TRIAL: NCT05599438
Title: Prospective, Longitudinal Study of 800 Recreational Athletes With Current and Former Use of Performance and Image Enhancing Drugs (PIED), Focusing on Androgenic Anabolic Steroids (AAS) - Rigshospitalet
Brief Title: Prospective, Longitudinal Study on FItness DOping in DenmarK
Acronym: FIDO-DK/RH
Status: Recruiting | Type: Observational
Sponsor: Caroline Michaela Kistorp (Other)
Collaborators: Copenhagen University Hospital at Herlev (Other); University Hospital Bispebjerg and Frederiksberg (Other); Centre for Preventative Doping Research at the German Sport University Cologne, Germany (Unknown); Body Identity Clinic, Odense, Denmark (Unknown)
Responsible Party: Sponsor-Investigator, Caroline Michaela Kistorp, Professor, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: H-21035759
Record Dates: First submitted 2022-10-19; First posted 2022-10-31 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Anabolic Steroid Overdose; Infertility; Cardiovascular Complication; Illicit Drug Use; Fitness; Mental Health Issue
Keywords: Cardiovascular Disease; Metabolic syndrome; Infertility; Mortality
MeSH Terms: conditions — Infertility; Cardiovascular Diseases; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Biospecimen Retention: Samples With DNA — Research biobank containing blood and urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Current users anabolic steroids: Current users of anabolic steroids with a use of more than 4 weeks
  Interventions: Other: No intervention
- Former users of anabolic steroids: Former users of anabolic steroids with a use of more than 4 weeks
  Interventions: Other: No intervention
- Healthy controls: 100 participants with no former use of anabolic steroids
  * 80 Male
  * 20 Female
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The aim of this prospective longitudinal study is to investigate the risks associated with use of anabolic steroids in fitness circles in Denmark in order to assess the scope of therapeutic need existing as a consequence of use. The objectives are:

* To assess long-term complications and outcomes related to: cardiovascular disease, diabetes, gonadal disease (women and men) and psychiatric disease using data from Danish registries including addressing central questions such as whether the following characteristics play a role for development of overt disease
* Characterization of illicit AAS use among men and women
* Current male reproductive health
* Current psychological well-being, aggressive tendencies, cognitive function and quality of life
* Current cardiovascular and metabolic status

The participants will undergo:

* Semi-structured medical interview
* Physical examinations
* Questionnaires
* Blood and urine sampling
* Dual X-ray Absorptiometry

With a subset undergoing further testing, including semen analysis, gonadotropin-releasing hormone (GnRH) and human chorionic gonadotropinm (hCG) stimulation and 82Rubidium positron emission tomography and computer tomography (PET/CT).

Register-based follow-up is planned every third year until the 15th year, marking the completion of the trial.

The study will include 800 participants with current or former AAS use and 100 participants (80 male; 20 female) as controls with no former or current use of AAS.

DETAILED DESCRIPTION:
Anabolic steroids (AAS) are synthetic derivates of the male sexhormone testosterone. The use of AAS is a growing phenomenon and have extended beyond the elite performance and body builder communities, involving a broader populace. The continued use causes a long-term impairment of testicular function, with symptoms of including impotence, depression, infertility and an increased risk of cardiovascular disease. AAS use is a clinical challenge as many psychological symptoms worsen in case of cessation of use. As AAS is often used by young individuals, the fulminant disease is rarely found by incidental screening. To assess long-term consequences, a large cohort is in need to be studied to accurately identify the risk of disease and when to initiate treatment. Furthermore, despite the use of AAS in women is present, the scientific community has thus far not taken notice, and the consequences are unknown, but are presumed to - beyond the changes in physical appearance - to include changes in fertility, risk of type 2 diabetes and cardiovascular disease. As AAS is acquired illicitly, the knowledge on the consequences of AAS use is sparse. No international or national consensus or recommendations exist as to the how to stop AAS use, screening of disease or therapeutic option in case of manifestations of symptoms or fulminant disease. The aim of the current study is to elucidate on the consequences of use of AAS in fitness circles in Denmark to assess the scope of therapeutic need.

ELIGIBILITY:
Inclusion Criteria:

- Male and female recreational athletes (≥18 years of age) with current or former illicit use (>3 months since AAS cessation) of PIEDs (e.g. AAS) for a minimum four weeks

Inclusion Criteria (Controls, n = 100):

- Male (n=80) or female (n=20) recreational athletes (≥18 years of age) with NO current or former illicit use of AAS.

Exclusion Criteria:

* Severe psychiatric or somatic diseases which makes it impossible to give informed consent or comply with the investigatory program.
* Known pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with current or former use of anabolic steroids of both male and female sex. The study also includes a control group (n=100 [male/female] - 80/20)
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2022-06-14 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2040-06-01 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular composite endpoint | 15 years
  Register-based composite of mortality, stroke, myocardial infarction, hospitalization due to heart failure and significant cardiovascular disease (See protocol)

SECONDARY OUTCOMES:
Fertility-related composite endpoint | 15 years
  Register-based composite of diagnoses related to fertility and testicular/ovarian function
Metabolism-related composite endpoint | 15 years
  Register-based composite of diagnosis related to impaired metabolic function (See protocol)
Mental health-related composite endpoint | 15 years
  Register-based composite of diagnosis related to psychiatric diagnosis (See protocol)
Male fertility | Baseline comparison when substudy is completed (expected 2023)
  Substudy analysis on difference in motile sperm count between groups (n=280 male participants; [current/former/controls] 60/60/80)
Myocardial flow reserve | Baseline comparison when substudy is completed (expected 2023)
  Substudy analysis on differences in myocardial flow reserve across groups (n=150 participants; male [current/former/controls]: 30/30/30; female [current/former/current]: 20/20/20)
hCG stimulation test | Baseline comparison when substudy is completed (expected 2023)
  Substudy analysis on difference in response to hCG stimulation test (n=60 male participants [former/controls]: 30/30)

OTHER OUTCOMES:
Anthropometry of the body composition of current and former users of AAS | Baseline comparison on entire cohort when initial completion is achieved (Date of primary completion)
  Analysis on group-differences in lean and fat mass evaluated by Dual X-ray Absorptiometry
Extensive examination of the mental health of current and former users of AAS using questionnaires | Baseline comparison on entire cohort when initial completion is achieved (Date of primary completion)
  Analysis on group-differences in response to questionnaires between current, former users of AAS and healthy controls (Questionnaires and further description found in protocol)
Extensive clinical characterization of current and former users of AAS | Baseline comparison on entire cohort when initial completion is achieved (Date of primary completion)
  Analysis on group-differences in clinical characteristics between current, former users of AAS and healthy controls (Measures and further description found in protocol)
Extensive biochemical profile of current and former users of AAS | Baseline comparison on entire cohort when initial completion is achieved (Date of primary completion)
  Analysis on group-differences in biochemical measures in blood and urine between current, former users of AAS and healthy controls (Measures and further description found in protocol)

CONTACTS AND LOCATIONS:
Overall Officials: Caroline M Kistorp, Professor, Principal Investigator — Centre for Cancer and Organ Disease, Department for Medical Endocrinology, Rigshospitalet
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
Due to national judicial restrictions individual participant data cannot be shared.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-30): https://cdn.clinicaltrials.gov/large-docs/38/NCT05599438/Prot_SAP_000.pdf